CLINICAL TRIAL: NCT00703118
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase III Trial of 2 Regimens of Telaprevir (With and Without Delayed Start) Combined With Pegylated Interferon Alfa-2a (Pegasys) and Ribavirin (Copegus) in Subjects With Chronic, Genotype 1, Hepatitis C Infection Who Failed Prior Standard Treatment
Brief Title: A Safety and Effectiveness Study of Telaprevir in Chronic, Genotype 1, Hepatitis C Patients That Failed Previous Standard Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tibotec BVBA (Industry)
Collaborators: Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR014842; VX-950-TIDP24-C216 (Other: Tibotec-Virco Virology BVBA)
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2013-12

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; Telaprevir; Peg-IFN-alfa-2a; Ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — telaprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A: T12/PR48 (Experimental): Participants will receive 12 weeks of 750 mg telaprevir eight hourly followed by 4 weeks of Placebo in combination with 48 weeks of Peg-IFN-alfa-2a and ribavirin at standard doses.
  Interventions: Drug: Telaprevir; Drug: Peg-IFN-alfa-2a; Drug: Ribavirin; Drug: Placebo
- Group B: T12(DS)/PR48 (Experimental): Participants will receive 4 weeks of Placebo followed by 12 weeks of 750 mg telaprevir eight hourly in combination with 48 weeks of Peg-IFN-alfa-2a and ribavirin at standard doses.
  Interventions: Drug: Telaprevir; Drug: Peg-IFN-alfa-2a; Drug: Ribavirin; Drug: Placebo
- Group C: Pbo/PR48 (Experimental): Participants will receive placebo in combination with Peg- IFN-alfa-2a and ribavirin for 16 weeks. Participants will receive Peg- IFN-alfa-2a and ribavirin for next 32 weeks.
  Interventions: Drug: Peg-IFN-alfa-2a; Drug: Ribavirin; Drug: Placebo

INTERVENTIONS:
Drug: Telaprevir — Participants will receive telaprevir tablets of 750 mg orally eight hourly for 12 weeks in group A and B.
  Arms: Group A: T12/PR48; Group B: T12(DS)/PR48
Drug: Peg-IFN-alfa-2a — Participants will receive 180 µg subcutaneous (under the skin) injection of Peg-IFN-alfa-2a once weekly for 48 weeks in Group A, B and C.
Drug: Ribavirin — Participants will receive ribavirin tablets of 1000-1200 mg orally twice daily for 48 weeks in Group A, B, and C.
Drug: Placebo — Participants will receive telaprevir matching placebo tablets orally for 4 weeks in Group A and B. Participants will receive telaprevir matching placebo tablets orally for 16 weeks in Group C.

SUMMARY:
The purpose of this study is to determine the safety, efficacy and tolerability of using two regimens of telaprevir (with and without delayed start) with standard treatment compared to standard treatment alone in participants with chronic, genotype 1, hepatitis C.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Phase III trial with telaprevir in patients with chronic Hepatitis C Virus (HCV), genotype 1, infection who failed prior treatment with standard treatment. Standard treatment is defined as treatment with Peg-INF and RBV. The trial is designed to compare the efficacy, safety, and tolerability of 2 regimens of telaprevir (with and without delayed start) combined with standard treatment versus standard treatment alone. The trial will consist of a screening period of approximately 4 weeks, a 48-week treatment period, and a 24-week follow-up period. Patients will be eligible to enroll in the trial if they (1) had an undetectable HCV Ribonucleic Acid (RNA) level at the end of a prior course of standard treatment but did not achieve a response (viral relapsers), or (2) never had an undetectable HCV RNA level during or at the end of a prior course of standard treatment (non-responders). Approximately 650 patients (350 prior relapsers and 300 prior non-responders) will be randomized in a 2:2:1 ratio to one of 3 treatment groups: Treatment group A will receive telaprevir with standard treatment for 12 weeks; followed by placebo with standard treatment for 4 weeks; followed by standard treatment for 32 weeks. Treatment group B will receive placebo with standard treatment for 4 weeks; followed by telaprevir with standard treatment for 12 weeks; followed by standard treatment for 32 weeks. Treatment group C will receive placebo with standard treatment for 16 weeks; followed by standard treatment for 32 weeks. In both telaprevir regimens (A and B), patients will receive 12 weeks of 750 mg of telaprevir every 8 hours along with 48 weeks of standard treatment. Telaprevir or placebo will be given by mouth at a dose of 750 mg every 8 hours for 16 weeks. Peg-INF will be given as an injection under the skin at a dose of 180 mcg once every week for 48 weeks. RBV will be given by mouth at a dose of either 1000 or 1200 mg (depending on your body weight) two times per day for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have chronic hepatitis C infection (genotype 1) with HCV RNA level >= 1000 IU/mL
* Patient must have failed at least 1 prior course of Peg-IFN/RBV therapy (standard treatment)
* Patient must be willing to use 2 effective methods of birth control for up to 7 months after last dose of study medication

Exclusion Criteria:

* Patient is a previous non-responder that is classified as a viral breakthrough case
* Patient is infected with Hepatitis C virus, genotype 1, exhibiting more than one subtype
* Patient has Hepatitis C virus, genotype 1, and exhibits co-infection with any other genotype
* Evidence of decompensated liver disease
* Patient has condition that requires use of systemic corticosteroids

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 663 (Actual)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA
Locations (91):
- United States (31):
  - Birmingham, Alabama
  - Coronado, California
  - La Jolla, California
  - Los Angeles, California
  - San Francisco, California
  - Aurora, Colorado
  - Bradenton, Florida
  - Gainesville, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Plymouth, Minnesota
  - Kansas City, Missouri
  - Egg Harbor Twp, New Jersey
  - Albuquerque, New Mexico
  - Manhasset, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Falls Church, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
- Australia (8):
  - Adelaide
  - Camperdown
  - Clayton
  - Darlinghurst
  - Kingswood
  - Melbourne
  - Parkville - Vic
  - Perth
- Austria (2):
  - Graz
  - Vienna
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- Brazil (4):
  - Distrito Barao Geraldo-Campina
  - Salvador
  - Santo André
  - São Paulo
- Canada (3):
  - Vancouver, British Columbia
  - Ottawa, Ontario
  - Montreal, Quebec
- France (9):
  - Clichy
  - Créteil
  - Grenoble
  - Lille
  - Lyon
  - Marseille
  - Paris
  - Pessac
  - Vandœuvre-lès-Nancy
- Germany (8):
  - Berlin
  - Cologne
  - Düsseldorf
  - Frankfurt
  - Freiburg im Breisgau
  - Hamburg
  - Hanover
  - München
- Israel (5):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Safed
  - Tel Aviv
- Netherlands (3):
  - Amsterdam-Zuidoost
  - Leiden
  - Nijmegen
- Poland (5):
  - Bialystok
  - Czeladź
  - Kielce
  - Lodz
  - Warsaw
- Santurce, Puerto Rico
- Spain (4):
  - Barcelona
  - Madrid
  - Seville
  - Valencia
- Stockholm, Sweden
- Switzerland (2):
  - Sankt Gallen
  - Zurich
- United Kingdom (2):
  - Birmingham
  - London

REFERENCES:
- [Derived] Zeuzem S, DeMasi R, Baldini A, Coate B, Luo D, Mrus J, Witek J. Risk factors predictive of anemia development during telaprevir plus peginterferon/ribavirin therapy in treatment-experienced patients. J Hepatol. 2014 Jun;60(6):1112-7. doi: 10.1016/j.jhep.2014.01.013. Epub 2014 Jan 29. PMID 24486089
- [Derived] Younossi Z, Negro F, Serfaty L, Pol S, Diago M, Zeuzem S, Andreone P, Lawitz EJ, Roberts S, Focaccia R, Foster GR, Horban A, Lonjon-Domanec I, Coate B, DeMasi R, Picchio G, Witek J. Homeostasis model assessment of insulin resistance does not seem to predict response to telaprevir in chronic hepatitis C in the REALIZE trial. Hepatology. 2013 Dec;58(6):1897-906. doi: 10.1002/hep.26437. Epub 2013 Oct 17. PMID 24382638
- [Derived] Pol S, Aerssens J, Zeuzem S, Andreone P, Lawitz EJ, Roberts S, Younossi Z, Foster GR, Focaccia R, Horban A, Pockros PJ, Van Heeswijk RP, De Meyer S, Luo D, Botfield M, Beumont M, Picchio G. Limited impact of IL28B genotype on response rates in telaprevir-treated patients with prior treatment failure. J Hepatol. 2013 May;58(5):883-9. doi: 10.1016/j.jhep.2012.12.023. Epub 2013 Jan 12. PMID 23321318
- [Derived] Zeuzem S, Andreone P, Pol S, Lawitz E, Diago M, Roberts S, Focaccia R, Younossi Z, Foster GR, Horban A, Ferenci P, Nevens F, Mullhaupt B, Pockros P, Terg R, Shouval D, van Hoek B, Weiland O, Van Heeswijk R, De Meyer S, Luo D, Boogaerts G, Polo R, Picchio G, Beumont M; REALIZE Study Team. Telaprevir for retreatment of HCV infection. N Engl J Med. 2011 Jun 23;364(25):2417-28. doi: 10.1056/NEJMoa1013086. PMID 21696308

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 105 sites in 17 countries: Argentina, Australia, Austria, Belgium, Brazil, Canada, Switzerland, Germany, Spain, France, United Kingdom, Israel, Italy, Netherlands, Poland, Sweden, and the United States.
Pre-assignment Details: 662 participants were treated (266 participants in the T12/PR48 group, 264 participants in the T12(DS)/PR48 group, and 132 participants in the Pbo/PR48 group) in this study.
Groups:
- T12/PR48: 12 weeks of 750 mg telaprevir eight hourly followed by 4 weeks of Placebo in combination with 48 weeks of Peg-IFN-alfa-2a and ribavirin at standard doses
- T12(DS)/PR48: 4 weeks of Placebo followed by 12 weeks of 750 mg telaprevir eight hourly in combination with 48 weeks of Peg-IFN-alfa-2a and ribavirin at standard doses
- Pbo/PR48: 48 weeks of Peg-IFN-alfa-2a and ribavirin at standard doses
Period: Overall Study
Arm/Group | T12/PR48 | T12(DS)/PR48 | Pbo/PR48
Started | 266 | 264 | 132
Completed | 245 | 248 | 110
Not Completed | 21 | 16 | 22
Not completed — Adverse Event | 1 | 2 | 2
Not completed — Subject Ineligible To Continue The Trial | 6 | 3 | 2
Not completed — Lost to Follow-up | 6 | 4 | 4
Not completed — Withdrawal by Subject | 8 | 7 | 13
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T12/PR48 | T12(DS)/PR48 | Pbo/PR48 | Total
Number analyzed (Participants) | 266 | 264 | 132 | 662
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (8.51) | 51 (8.24) | 49.9 (9.74) | 50.6 (8.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 75 | 44 | 202
  Male | 183 | 189 | 88 | 460
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 6 | 2 | 3 | 11
  Black or African American | 11 | 8 | 11 | 30
  White | 246 | 252 | 117 | 615
  Other | 3 | 2 | 1 | 6
AgeCategoricalOther [Number; unit: participants]
  >= 45 years | 64 | 55 | 40 | 159
  Between 45 and 65 years | 197 | 201 | 85 | 483
  >= 65 years | 5 | 8 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Virologic Response (SVR) 24 Weeks After the Last Planned Dose of Study Medication - SVR24 Planned
Description: SVR24 planned is defined as having undetectable plasma Hepatitis C virus (HCV) ribonucleic acid (RNA) levels 24 weeks after the last planned dose of study medication.
Time Frame: Week 72
Population: Full Analysis Set: All randomized participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | T12/PR48 | T12(DS)/PR48 | Pbo/PR48
Number analyzed (Participants) | 266 | 264 | 132
Participants | 171 | 175 | 22
Statistical Analysis 1: Comparison: T12/PR48 vs Pbo/PR48; Null hypothesis: Assuming a 55% response rate in the groups receiving Treatment T12/PR48, a 29% response rate in the group receiving Treatment Pbo/PR48, a 2-sided continuity corrected Chi-squared test, with an overall significance level of 5% and a 2:2:1 randomization, a sample size of 140 patients receiving Treatment T12/PR48 and 70 patients in receiving Treatment Pbo/PR48 provided a power of approximately 90% to demonstrate a statistically significant difference; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Overall significance level was set at 5% (two-sided). Adjustment of significance level for multiple comparisons was carried out using the Hochberg procedure; Included: treatment, type of prior response (relapser, partial responder, null-responder) and their interaction, and baseline HCV RNA as a covariate; Difference in percentage of response = 46.8, 95% CI 2-sided [36.8 to 56.7] — Difference in percentage of response was estimated through the logistic regression model
Statistical Analysis 2: Comparison: T12(DS)/PR48 vs Pbo/PR48; Null hypothesis: Assuming a 55% response rate in the groups receiving Treatment T12/PR48 or T12(DS)/PR48, a 29% response rate in the group receiving Treatment Pbo/PR48, a 2-sided continuity corrected Chi-squared test, with an overall significance level of 5% and a 2:2:1 randomization, a sample size of 140 patients receiving Treatment T12(DS)/PR48 and 70 patients in receiving Treatment Pbo/PR48 provided a power of approximately 90% to demonstrate a statistically significant difference; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in percentage of response = 49.8, 95% CI 2-sided [39.9 to 59.7] — Difference in percentage of response was estimated through the logistic regression model

2. Secondary Outcome: Number of Participants Acheiving Rapid Virologic Response (RVR) at Week 4
Description: RVR was defined as having undetectable Hepatitis C virus (HCV) ribonucleic acid (RNA) at Week 4.
Time Frame: Week 4
Population: All analyses were performed on the full analysis (FA) set, which was defined as all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | T12/PR48 | T12(DS)/PR48 | Pbo/PR48
Number analyzed (Participants) | 266 | 264 | 132
Participants | 152 | 188 | 3

3. Secondary Outcome: Number of Participants Acheiving Undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels at Week 48 (End of Treatment)
Time Frame: Week 48
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | T12/PR48 | T12(DS)/PR48 | Pbo/PR48
Number analyzed (Participants) | 266 | 264 | 132
Participants | 184 | 191 | 49

4. Secondary Outcome: Number of Participants With Sustained Virologic Response (SVR) 12 Weeks After the Last Planned Dose of Study Medication - SVR12 Planned
Description: SVR12 planned was defined as having undetectable plasma Hepatitis C virus (HCV) ribonucleic acid (RNA) levels 12 weeks after the last planned dose of study medication (SVR12 planned).
Time Frame: Week 60
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | T12/PR48 | T12(DS)/PR48 | Pbo/PR48
Number analyzed (Participants) | 266 | 264 | 132
Participants | 175 | 178 | 22

5. Secondary Outcome: Number of Participants Who Meet the Telaprevir Stopping Rule at Week 4, Week 6, or Week 8
Description: Telaprevir stopping rule is defined as having Hepatitis C virus (HCV) ribonucleic acid (RNA) levels >100 IU/mL at Week 4, Week 6, or Week 8 after start of telaprevir.
Time Frame: Week 4, Week 6, or Week 8
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | T12/PR48 | T12(DS)/PR48
Number analyzed (Participants) | 266 | 264
Participants
  Week 4 | 16 | 14
  Week 6 | 5 | 2
  Week 8 | 2 | 0

6. Secondary Outcome: Number of Participants Who Have Viral Relapse During Entire Follow-up Period (up to Week 72)
Description: Viral relapse was defined as having confirmed detectable Hepatitis C virus (HCV) ribonucleic acid (RNA) levels during entire follow-up period (up to Week 72).
Time Frame: Up to Week 72
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | T12/PR48 | T12(DS)/PR48 | Pbo/PR48
Number analyzed (Participants) | 266 | 264 | 132
Participants | 26 | 27 | 33

7. Secondary Outcome: Change From Baseline in log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Week 4
Time Frame: Baseline (Day 1) to Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | T12/PR48 | T12(DS)/PR48 | Pbo/PR48
Number analyzed (Participants) | 245 | 240 | 121
log10 IU/mL | -5.5 (1.06) | -2.0 (1.42) | -1.9 (1.40)

8. Secondary Outcome: Number of Participants Acheiving Extended Rapid Virologic Response at Week 4 and Week 12
Description: Extended rapid virologic response was defined as undetectable Hepatitis C virus (HCV) ribonucleic acid (RNA) levels.
Time Frame: Week 4 and Week 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | T12/PR48 | T12(DS)/PR48 | Pbo/PR48
Number analyzed (Participants) | 266 | 264 | 132
Participants | 141 | 180 | 3

ADVERSE EVENTS:
Time Frame: 72 weeks
Groups:
- T12/PR48 - TVR/PBO TREATMENT: 12 weeks of 750 mg telaprevir q8hr followed by 4 weeks of Placebo in combination with 48 weeks of Peg-IFN-alfa-2a and RBV at standard doses - TE AEs during the telaprevir/placebo treatment phase
- T12(DS)/PR48 - TVR/PBO TREATMENT: 4 weeks of Placebo followed by 12 weeks of 750 mg telaprevir q8hr in combination with 48 weeks of Peg-IFN-alfa-2a and RBV at standard doses - TE AEs during the telaprevir/placebo treatment phase
- Pbo/PR48 - TVR/PBO TREATMENT: 48 weeks of Peg-IFN-alfa-2a and RBV at standard doses - TE AEs during the telaprevir/placebo treatment phase
- T12/PR48 - OVERALL TREATMENT: 12 weeks of 750 mg telaprevir q8hr followed by 4 weeks of Placebo in combination with 48 weeks of Peg-IFN-alfa-2a and RBV at standard doses - TE AES during the overall treatment phase
- T12(DS)/PR48 - OVERALL TREATMENT: 4 weeks of Placebo followed by 12 weeks of 750 mg telaprevir q8hr in combination with 48 weeks of Peg-IFN-alfa-2a and RBV at standard doses - TE AES during the overall treatment phase
- Pbo/PR48 - OVERALL TREATMENT: 48 weeks of Peg-IFN-alfa-2a and RBV at standard doses - TE AEs during the overall treatment phase
Arm/Group | T12/PR48 - TVR/PBO TREATMENT | T12(DS)/PR48 - TVR/PBO TREATMENT | Pbo/PR48 - TVR/PBO TREATMENT | T12/PR48 - OVERALL TREATMENT | T12(DS)/PR48 - OVERALL TREATMENT | Pbo/PR48 - OVERALL TREATMENT
Serious Adverse Events (participants affected / at risk) | 18/266 | 17/264 | 4/132 | 33/266 | 32/264 | 7/132
Other Adverse Events (participants affected / at risk) | 253/266 | 255/264 | 126/132 | 257/266 | 260/264 | 126/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T12/PR48 - TVR/PBO TREATMENT (N=266) | T12(DS)/PR48 - TVR/PBO TREATMENT (N=264) | Pbo/PR48 - TVR/PBO TREATMENT (N=132) | T12/PR48 - OVERALL TREATMENT (N=266) | T12(DS)/PR48 - OVERALL TREATMENT (N=264) | Pbo/PR48 - OVERALL TREATMENT (N=132)
Anaemia (Blood and lymphatic system disorders) | 4 | 5 | 1 | 6 | 7 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 3 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 1
Cardiac valve disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Basedow's disease (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Caecitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Multiple drug overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Blood corticotrophin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 2 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Cerebral thrombosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Coma (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0
Substance abuse (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 2 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T12/PR48 - TVR/PBO TREATMENT (N=266) | T12(DS)/PR48 - TVR/PBO TREATMENT (N=264) | Pbo/PR48 - TVR/PBO TREATMENT (N=132) | T12/PR48 - OVERALL TREATMENT (N=266) | T12(DS)/PR48 - OVERALL TREATMENT (N=264) | Pbo/PR48 - OVERALL TREATMENT (N=132)
Anaemia (Blood and lymphatic system disorders) | 70 | 82 | 17 | 78 | 93 | 19
Leukopenia (Blood and lymphatic system disorders) | 23 | 13 | 9 | 27 | 20 | 11
Neutropenia (Blood and lymphatic system disorders) | 17 | 24 | 12 | 38 | 35 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 14 | 6 | 9 | 16 | 7
Vision blurred (Eye disorders) | 10 | 7 | 2 | 16 | 10 | 3
Abdominal pain (Gastrointestinal disorders) | 32 | 29 | 16 | 43 | 36 | 21
Anal pruritus (Gastrointestinal disorders) | 14 | 15 | 0 | 14 | 15 | 0
Anorectal discomfort (Gastrointestinal disorders) | 20 | 11 | 0 | 21 | 11 | 0
Constipation (Gastrointestinal disorders) | 11 | 11 | 5 | 20 | 17 | 5
Diarrhoea (Gastrointestinal disorders) | 60 | 64 | 16 | 66 | 69 | 18
Dry mouth (Gastrointestinal disorders) | 23 | 20 | 12 | 25 | 21 | 12
Dyspepsia (Gastrointestinal disorders) | 13 | 15 | 10 | 13 | 18 | 11
Haemorrhoids (Gastrointestinal disorders) | 38 | 28 | 7 | 40 | 32 | 9
Nausea (Gastrointestinal disorders) | 89 | 80 | 31 | 94 | 87 | 31
Vomiting (Gastrointestinal disorders) | 29 | 28 | 10 | 37 | 31 | 11
Asthenia (General disorders) | 49 | 55 | 35 | 51 | 60 | 38
Chills (General disorders) | 41 | 31 | 19 | 42 | 31 | 19
Fatigue (General disorders) | 138 | 124 | 51 | 145 | 131 | 53
Influenza like illness (General disorders) | 85 | 90 | 33 | 85 | 94 | 33
Injection site erythema (Injury, poisoning and procedural complications) | 14 | 19 | 5 | 15 | 20 | 6
Irritability (General disorders) | 31 | 36 | 19 | 36 | 38 | 21
Pain (General disorders) | 14 | 5 | 3 | 16 | 5 | 4
Pyrexia (General disorders) | 57 | 63 | 32 | 59 | 71 | 36
Nasopharyngitis (Infections and infestations) | 6 | 10 | 7 | 8 | 11 | 8
Weight decreased (Investigations) | 7 | 5 | 6 | 12 | 18 | 7
Anorexia (Metabolism and nutrition disorders) | 32 | 33 | 19 | 33 | 36 | 19
Decreased appetite (Metabolism and nutrition disorders) | 16 | 19 | 7 | 17 | 23 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 27 | 19 | 36 | 31 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 14 | 8 | 25 | 21 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 6 | 4 | 14 | 10 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 35 | 40 | 24 | 45 | 42 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 7 | 2 | 15 | 12 | 2
Disturbance in attention (Nervous system disorders) | 5 | 13 | 8 | 7 | 17 | 9
Dizziness (Nervous system disorders) | 18 | 23 | 5 | 19 | 27 | 7
Dysgeusia (Nervous system disorders) | 32 | 27 | 8 | 33 | 32 | 8
Headache (Nervous system disorders) | 106 | 101 | 46 | 112 | 109 | 49
Anxiety (Psychiatric disorders) | 6 | 21 | 11 | 9 | 26 | 13
Depression (Psychiatric disorders) | 20 | 33 | 14 | 24 | 35 | 19
Insomnia (Psychiatric disorders) | 55 | 70 | 29 | 68 | 84 | 34
Sleep disorder (Psychiatric disorders) | 10 | 8 | 7 | 11 | 11 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 44 | 49 | 23 | 62 | 66 | 26
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 | 41 | 16 | 32 | 50 | 17
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 11 | 17 | 5 | 15 | 20 | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 12 | 5 | 13 | 18 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 19 | 12 | 38 | 40 | 17
Dry skin (Skin and subcutaneous tissue disorders) | 36 | 45 | 21 | 44 | 53 | 21
Erythema (Skin and subcutaneous tissue disorders) | 19 | 15 | 5 | 27 | 16 | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 9 | 6 | 6 | 9 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 132 | 130 | 35 | 138 | 132 | 36
Rash (Skin and subcutaneous tissue disorders) | 91 | 88 | 24 | 99 | 95 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days